CLINICAL TRIAL: NCT06628180
Title: Investigation of Accelerated LIFU: Towards Therapeutic Use for Chronic Pain
Brief Title: LIFU for Chronic Pain
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Collaborators: Focused Ultrasound Foundation (Other)
Responsible Party: Principal Investigator, Wynn Legon, Assistant Professor, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 24-994
Record Dates: First submitted 2024-09-24; First posted 2024-10-04 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Chronic Pain
Keywords: low-intensity focused ultrasound; LIFU; tFUS
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Sham LIFU (Sham Comparator): Sham application of LIFU - all follow up (MRI, questionnaires) will be identical.
  Interventions: Device: Sham LIFU
- Verum LIFU (Experimental): Active LIFU application with 3 week follow-up (MRI, questionnaires)
  Interventions: Device: LIFU

INTERVENTIONS:
Device: LIFU — Application of low-intensity focused ultrasound for neuromodulation
  Arms: Verum LIFU
Device: Sham LIFU — Sham application of LIFU - will appear the same to participants.
  Arms: Sham LIFU

SUMMARY:
This research project is examining the effects of noninvasive brain stimulation on chronic pain. We believe this study will help us to better understand possible treatments for chronic pain patients. Subjects will undergo functional magnetic resonance imaging (fMRI) and a computed tomography (CT) scan, which is a way to take pictures of the brain and skull. Subjects will receive noninvasive brain stimulation using low-intensity focused ultrasound (LIFU) sound waves, to temporarily change brain activity. Subjects will undergo pain testing using a small device that will increase the temperature of their skin and will rate this pain. Brain signals (EEG), heart rate and rhythm, blood pressure, respiration rate, and skin moisture will be monitored. Subjects will complete behavioral questionnaires. Each study session is expected to take 1.5-3 hours. Total participation takes 10 weeks.

DETAILED DESCRIPTION:
This is a 2-arm, sham-controlled, cross-over design. This study is collected over 5-7 study visits.

Initial Imaging (1): MRI and CT scans, Questionnaires, and QST Testing.

Intervention (2): Sham or verum LIFU application every 10 minutes, totaling in 8 applications. Between LIFU or Sham application quantitative sensory testing (QST) will be performed. Physiological data collection such as EEG, EDA, BP, ECG, and Respiration will be collected throughout the study visit.

Follow-Up Imaging (2-4): Following intervention sessions participants will receive a resting-state MRI. This can occur throughout the 4-weeks following an intervention visit. Participants will be scanned at least once after each intervention session.

Follow-Up Virtual Questionnaires: Following intervention sessions participants will receive a link (or a phone call if preferred) to periodically rate their pain and report on various lifestyle impacts of their chronic pain. Participants will complete these questionnaires at least twice per week in the 2 weeks following an intervention visit. These questionnaires will take less than 30 minutes.

After completing the intervention and minimum 4-week washout period, the participant will return for a second intervention visit and 3 week follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a chronic pain diagnosis. Pain must be moderate-to-severe and present for at least 3 months prior to research participation. Patients of all ethnicities, who understand and speak English.

Exclusion Criteria:

* Claustrophobia (scanning environment may be uncomfortable).
* Contraindications to MRI: including pacemaker, aneurysm clips, neurostimulators, cochlear implants, metal in eyes, steel worker, or other implants.
* Contraindications to CT: pregnancy
* Active medical disorder or treatment with potential CNS effects (e.g. Alzheimer's)
* History of neurologic disorder. (e.g. Parkinson's, Epilepsy, or Essential Tremor)
* History of head injury resulting in loss of consciousness for >10 minutes.
* History of alcohol or drug dependence (through self-report).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-01-30 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Pain sensation | during 2 study visits - up to 8 times per visit.
  Reduced perceived sensation (pain) score in response to painful stimulus. Pain scale of 0-10, 0 being no pain and 10 being worst pain imaginable.

SECONDARY OUTCOMES:
Quality of Life | 4 weeks following each intervention, every 2-4 days, 30 min per day.
  quality of life questionnaires over a 4 week period following intervention

OTHER OUTCOMES:
rs-fMRI | pre and post intervention, up to 5 scans (1 pre, up to 4 post)
  Changes in resting state functional connectivity.

CONTACTS AND LOCATIONS:
Locations (1):
- Fralin Biomedical Research Institute at VTC, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: No